CLINICAL TRIAL: NCT05024461
Title: Comparison of the Results, Feasibility and Acceptability of Molecular Detection of SARS-CoV2 Between Nasopharyngeal Swab Specimens Recovered in Virological Transport Medium and Those Obtained by Salivary Sputum
Brief Title: Comparison of Detection of SARS-CoV2 (COVID-19) Between Nasopharyngeal Swab Specimens and Those Obtained by Salivary Sputum
Acronym: COVISAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVISAL
Record Dates: First submitted 2021-08-16; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with an indication for a COVID19 test (Experimental): The persons included will be those who have an indication for a COVID 19 test and who present themselves at the Cayenne hospital and during the screening missions organised by the Red Cross and Médecin du Monde during the COVID 19 epidemic in the territory
  Interventions: Diagnostic Test: Salivary test for COVID19

INTERVENTIONS:
Diagnostic Test: Salivary test for COVID19 — Results of nasopharyngeal and salivary samples taken at the Cayenne hospital and the Caen university center,
  * Pre-analytical particularities and analytical particularities
  * Cycle threeshold
  * Demographic variables
  * Clinical variables
  * Clinical criteria
  * Questionnaire on the perception of the 2 sampling methods

SUMMARY:
Multicenter observational study of diagnostic test validation (Research Involving the Human Person, type 3) In addition to the diagnosis by the reference method (nasopharyngeal swab), the patient will be asked to provide a saliva sample via a salivary spit. The clinical circumstances of the diagnosis, the age of the patient, the associated terrain (diabetes, immunodepression, pregnancy) will be noted. The nasopharyngeal and saliva samples will be analyzed in Cayenne and the remaining samples will be frozen and stored at the CRB before being sent to the University Hospital of Caen for analysis and concordance verification.

The expected benefits are:

Possibility of repeating tests in the same person more easily due to the absence of pain and thus reduce the barriers to diagnosis and screening.

Possibility of self-sampling, which could simply be sent to the laboratory, which would relieve the diagnostic sites that mobilize staff and require a fairly heavy organization. Avoid long waiting lines that can be an obstacle and lead to a renunciation of the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an indication to perform a COVID diagnostic test (symptomatology, contact case, systematic screening etc...)
* Men and women at least 3 years old

Exclusion Criteria:

* Refusal of the patient or his legal representative,
* Taking treatments that reduce salivary volume (anticholinergic activity)
* Impossibility to perform the nasopharyngeal test
* Patient under guardianship or curatorship, persons placed under protective measures

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1159 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2021-11-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of salivary test vs. nasopharyngeal test | 1 day

SECONDARY OUTCOMES:
- Proportion of analyses not performed on salivary samples for the following reasons (vs. number of salivary sample analyses performed): o Insufficient quantity of biological sample, o Inability to collect the sample | 1 day
Perception of the tests by questionnaire (proportion of positive opinions) | 1 day
Perception of the tests by questionnaire (proportion of negative opinions) | 1 day
Positivity and negativity of the salivary test vs. symptomatology and associated terrain | 1 day
Sensitivity and specificity analysis between the salivary test and the nasopharyngeal test according to the clinical context | 1 day
  Sensitivity and specificity analysis between the salivary test and the nasopharyngeal test according to the time between the samples and the onset of symptoms, the time between the samples and the contact with an index case, the known immunodepression and the clinical context (diabetes, pregnancy)
Description of the aspect of the saliva collected: mucous or fluid | 1 day
  Description of the analytical criteria of the saliva sample
Volume of saliva collected (mL) | 1 day
  Description of the analytical criteria of the saliva sample: (pipette measurement, if the saliva is not fluid, pipette measurement after vortexing for 1 min)
Description of the analytical criteria of the saliva sample:pre-analytical treatments if necessary | 1 day
Number of Cycle threeshold for the first analysis (done at the Cayenne hospital) and the second analysis (done at the university hospital of Caen) | 1 day
- Sensitivity of salivary test vs nasopharyngeal test with strong positives (3 genes detected) | 1 day
- Specificity of salivary test vs nasopharyngeal test with strong positives (3 genes detected) | 1 day
- Sensitivity of salivary test vs nasopharyngeal test with weak positives (1 gene detected) | 1 day
- Specificity of salivary test vs nasopharyngeal test with weak positives (1 gene detected) | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Cayenne, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: No